CLINICAL TRIAL: NCT00820144
Title: Functional Exploration of the Immune Response Using the B-Subunit of Cholera Toxin Administered by Mucosal Way in Healthy Adult Volunteer: Potential Role in Development of Vaccine Processes
Brief Title: Cholera Toxin B Subunit (CTB) Administered by Mucosal Way in Healthy Adult Volunteer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Departement de la recherche Clinique et de l'Innovation, CHU de NICE
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: PHRC 2003 CTB
Record Dates: First submitted 2009-01-02; First posted 2009-01-12 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Infection
Keywords: immune response; b-subunit of cholera toxin; mucosal way; healthy volonteers; vaccine
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): voie nasale 0.25 mg
  Interventions: Biological: CTB by nasal way
- 2 (Experimental): 0.5mg of CTB by oral way
  Interventions: Biological: absorption of CTB by oral way
- 3 (Experimental): 1mg of dukoral by oral way
  Interventions: Biological: absorption of dukoral by oral way
- 4 (Experimental): 0.25mg of CTB by sublingual way
  Interventions: Biological: absorption of CTB by sublingual way
- 5 (Experimental): 1mg of CTB by sublingual way
  Interventions: Biological: absorption of CTB by sublingual way

INTERVENTIONS:
Biological: CTB by nasal way
  Arms: 1
Biological: absorption of CTB by oral way — absorption of CTB by oral way
  Arms: 2
Biological: absorption of dukoral by oral way — absorption of dukoral by oral way
  Arms: 3
Biological: absorption of CTB by sublingual way — absorption of CTB by sublingual way
  Arms: 4
Biological: absorption of CTB by sublingual way — absorption of CTB by sublingual way
  Arms: 5

SUMMARY:
It is a biomedical research without direct individual benefit, exploring and comparing the mucosal immune response after oral, nasal and sublingual administration of B-subunit of non-toxic cholera toxin (CTB) in healthy adult volunteers.

DETAILED DESCRIPTION:
The immense majority of the infections involve the mucosal surfaces as a gateway of the pathogenic agent. These mucosal surfaces are mainly represented by the gastrointestinal, respiratory and urogenital tract. These mucosal surfaces contain a highly developed immune system, which can exploit in a mucus vaccine approach to fight against infectious agents upon their penetration in the body. It has been established that to be effective against infection mucosa, a vaccine must stimulate the local immune system. This objective is reached much more efficiently when the vaccine is administered by mucosal way (oral, nasal) than by the parenteral classical way. Recent works allowed developing a new non invasive system of administration of vaccines. It is based on the mucosal administration (oral, nasal, rectal, vaginal) comprising a combination of antigen bound (either chemically or by genetic fusion) to the non-toxic subunit of cholera toxin or CTB (Cholera Toxin B subunit). This subunit has an exceptional affinity for GM1 ganglioside expressed on the surface of all nucleated cells. So, the mucosal administration (by oral or nasal route) of a low dose of an antigen linked to the CTB - Mucosal vector with immunomodulatory properties - Leads powerful secretor immune responses in the exposed mucous As well as in distant mucous, with a strong production of secretories IgA.

The developed methods of exploration have to allow to characterize the cells which live (or which migrate) in the mucous membrane investigated on the functional and phenotypic plan.

This research should lead to a range of standardized operating procedures, allowing to evaluate the immunogenicity of vaccines candidates to the mucous administration and of predictive markers of the type of immune response generated.

The main objective of the study is to analyse at the healthy voluntary subjects the systematic immunizing answer induced after nasal, oral or sublingual administration of the CTB from blood samples - the lymphoid "compartment" the most accessible at the man- from saliva and from nasal wash. The immune response after administration of the CTB By sublingual way should be comparable in that of two other ways in term of intensity of the response, however, with a different IgA / IgG report.

The secondary objective of the study is to establish a range of tests to predict the character and the intensity of this response by analyzing the expression of B cells certain surface molecules marking their future for the production of Antibodies.

It is a regional prospective monocentric study conducted in opened without direct individual profit. The study will be conducted over 3 years including 24 months of recruitment for each patient with a follow-up of 35 days and 6 months of operation data.

ELIGIBILITY:
Inclusion Criteria:

* Adult male between 18 and 50 years,
* Adult female aged 18 to 50 years under oral contraception (pill) for at least 6 months, or IUD for at least 6 under, and agreeing to carry out a pregnancy test during the initial clinical visit
* Affiliate or entitled to Social Security
* Signing the informed consent of the volunteer

Exclusion Criteria:

* Seropositive patient for HIV, Hepatitis B, Hepatitis C (oral questioning)
* Pregnant Woman, parturient or breast-feeding
* News hospitalized for other reasons that the research
* Minor, Major under supervision
* Participation in a current or recent study or at present in period of exclusion

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2006-04; Primary Completion 2006-04 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The primary criteria which will estimate this immune response is the production of immunoglobulin A1, A2 and G totals specific to the CTB contained at the level of salivary secretions or produced by mononuclear cells of peripheral blood. | every week during 5 weeks

SECONDARY OUTCOMES:
The secondary criteria of judgment are other phenotypic and functional changes induced on the immune cells present in saliva or in the blood after administration of CTB. | every week during 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul HOFMAN, Professor, Principal Investigator — Departement d'anatomo-pathologie, CHU de Nice
Locations (1):
- Laboratoire d'anatomo-pathologie, hôpital Pasteur, Nice, France